CLINICAL TRIAL: NCT03624725
Title: A Single-center, Randomized, Controlled Clinical Study of the Effects of Modified and Traditional BII+Braun Digestive Tract Reconstruction Methods on Quality of Life After Radical Gastrectomy for Distal Gastric Cancer
Brief Title: A Clinical Study of the Effects of Modified BII+Braun on Quality of Life After for Distal Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xue Yingwei (Other)
Responsible Party: Sponsor-Investigator, Xue Yingwei, Director, Head of Gastrointestinal surgery, Principal Investigator, Clinical Professor, The Third Affiliated Hospital of Harbin Medical University
Organization: The Third Affiliated Hospital of Harbin Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-02-R
Record Dates: First submitted 2018-07-29; First posted 2018-08-10 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Quality of Life
Keywords: Gastric cancer; Quality of life
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified BII+Braun (Active Comparator): The jejunum of the input segment is properly ligated with double line 7 at 3-5cm from the anastomotic site, and the jejunum of the output segment is extended to 30cm
  Interventions: Procedure: modified BII+Braun
- traditional BII+Braun (No Intervention): traditional BII+Braun digestive tract reconstruct

INTERVENTIONS:
Procedure: modified BII+Braun — modified BII+Braun digestive tract reconstruction
  Arms: modified BII+Braun

SUMMARY:
The jejunum of the input segment is properly ligated with double line 7 at 3-5cm from the anastomotic site, and the jejunum of the output segment is extended to 30cm

DETAILED DESCRIPTION:
The T1-4a N0-3 M0 gastric adenocarcinoma patients were used to evaluate whether the quality of life after modified BII+Braun digestive tract reconstruction was superior to the traditional BII+Braun digestive tract reconstruction

ELIGIBILITY:
Inclusion Criteria:

* 18<age<75
* Gastric lesions were diagnosed as gastric adenocarcinoma by endoscopic biopsy
* The preoperative clinical stage is T1-4a,N0-3,M0(According to AJCC- 7th TNM tumor stage)
* It is expected that the results of R0 surgery can be obtained by performing distal gastrectomy and D2 lymph node dissection
* Preoperative ECOG performance status score 0/1
* Nutrition risk screening（NRS2002）
* Preoperative ASA score I-III
* Patient informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding women
* Severe mental illness
* History of upper abdominal surgery
* History of gastric surgery (including ESD/EMR for gastric cancer)
* 3 years of history of other malignant diseases；
* Gastric cancer patients who have undergone neoadjuvant treatment or recommend neoadjuvant treatment
* A history of unstable angina or myocardial infarction within 6 months
* History of cerebral infarction or cerebral hemorrhage within 6 months
* There is a history of sustained systemic corticosteroid treatment within 1 month
* Needs simultaneous surgical treatment of other diseases；
* Gastric cancer complications (bleeding, perforation, obstruction) require emergency surgery
* Pulmonary function test FEV<1 predicted value 50%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Effects of quality of life | The quality of life questionnaire was conducted at six months after surgery.
  The GSRS scoring system was used to understand the functional status of the digestive tract and its impact on quality of life in postoperative patients .The GSRS scoring system was 0-3, with 0 being the mildest and 3 being the most severe

CONTACTS AND LOCATIONS:
Overall Officials: Yingwei Xue, doctor, Study Director — Director of Gastrointestinal surgery
Locations (1):
- Gastrointestinal surgery of the affiated tumor hospital, Harbin, Helongjiang, China

REFERENCES:
- [Derived] Cai Z, Mu M, Ma Q, Liu C, Jiang Z, Liu B, Ji G, Zhang B. Uncut Roux-en-Y reconstruction after distal gastrectomy for gastric cancer. Cochrane Database Syst Rev. 2024 Feb 29;2(2):CD015014. doi: 10.1002/14651858.CD015014.pub2. PMID 38421211